CLINICAL TRIAL: NCT00312182
Title: Evaluation Of The Effect Of Nelfinavir On QT Intervals At Steady-State After Twice-Daily Administration Of Nelfinavir Tablets To Healthy Volunteers
Brief Title: Thorough QT Study of Nelfinavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A4301023
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir

SUMMARY:
To assess if nelfinavir has any clinically meaninful effect on cardiac function, namely ECG evaluation

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 and 55 years, inclusive. Body Mass Index (BMI) of approximately 18 to 30 kg/m2.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2006-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
ECG evaluation

SECONDARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (2):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Ann Arbor, Michigan
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4301023&StudyName=Thorough+QT+study+of+Nelfinavir